CLINICAL TRIAL: NCT05667181
Title: The Application Value of da Vinci Linear Cutting Stapler SureForm in Robotic Anus Preserving Surgery for Rectal Cancer: a Single Center Prospective Randomized Controlled Trial
Brief Title: The Application Value of da Vinci Linear Cutting Stapler SureForm in Robotic Anus Preserving Surgery for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchang University (Other)
Responsible Party: Principal Investigator, Taiyuan Li, professor, Nanchang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022155
Record Dates: First submitted 2022-12-10; First posted 2022-12-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Rectal Cancer; Robotic; Anastomotic Leak; Laparoscopic
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- robotic group (Experimental): Robot linear cutting stapler
  Interventions: Device: Surform
- laparocaopic group (Active Comparator): laparoscopic linear cutting stapler
  Interventions: Device: Surform

INTERVENTIONS:
Device: Surform — Da Vinci linear cutting stapler

SUMMARY:
Anastomotic complications are serious complications after anus preserving surgery for rectal cancer,the instrument anastomosis technology are one of the factors that influence the occurrence of anastomotic complications after surgery,the laparoscopic linear cutting closure device used in robotic rectal cancer may increase the occurrence of anastomotic complications,but the robot linear cutting stapler (SureForm) may reduce the incidence of postoperative anastomotic complications due to the technical advantages,therefore,the aim of this study is to evaluate the impact of robotic linear cutting stapler SureForm and laparoscopic linear cutting stapler on the incidence of anastomotic complications after robotic rectal cancer anus preserving surgery.

DETAILED DESCRIPTION:
Anastomotic complications are serious complications after anus preserving surgery for rectal cancer, including anastomotic leakage, anastomotic bleeding, and anastomotic stenosis, with a incidence rate of 1.6% - 20.5% . The occurrence of anastomotic complications increases the perioperative mortality, hospital stay, and hospital costs of patients, and even some patients with severe anastomotic complications need to be re operated after surgery, which seriously affects the quality of life of patients. More research shows that , The complications of anastomotic stoma lead to the delay of postoperative adjuvant therapy, which increases the local recurrence rate of tumor. Therefore, how to reduce the occurrence of anastomotic complications in anus preserving surgery for rectal cancer has always been the focus of surgeons.

A variety of factors are involved in the occurrence of anastomotic complications after surgery, including gender, patient's general condition, tumor size and distance from anal margin, and instrument anastomosis technology . It is believed that , when using a closer to break the rectum during radical resection of rectal cancer, the use of multiple nail cages will increase the incidence of postoperative anastomotic complications. In the past, laparoscopic rectal cutting staplers were used in robotic radical resection of rectal cancer, and most of them were completed with the cooperation of assistants. In difficult cases, the mechanical arm needed to be removed and the main knife was used to perform rectal resection. In addition, the laparoscopic linear cutting closure device was cumbersome and complicated, and it often needed to use multiple nail silos to cut rectum in a narrow pelvic cavity, resulting in uneven anastomosis quality, Increase the occurrence of anastomotic complications. In recent years, the robot company has developed a new software driven robot assisted stapler (SureForm). The stapler can be directly loaded onto the mechanical arm. When the rectum is broken, the main knife can independently control it on the console. It has a joint head that rotates 60 ° from top to bottom, left to right, a 120 ° cone range of motion, and a 540 ° wrist joint design of the rod body, so that the stapler jaws can be vertically placed and separated from the rectum, The utility model can reduce the use of the nail bin when the rectum is transected, thereby reducing the incidence of postoperative anastomotic complications.

At present, only a few foreign studies have reported the application of robot linear cutting stapler SureForm in anus preserving surgery for rectal cancer, and the studies are retrospective, with a small sample size. There is no report in China. Therefore, this study adopts a prospective randomized controlled study method to evaluate the impact of robotic linear cutting stapler SureForm and laparoscopic linear cutting stapler on the incidence of anastomotic complications after robotic rectal cancer anus preserving surgery, so as to provide a reference for the application of robotic linear cutting stapler SureForm in robotic anus preserving surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The age is more than 18 years old and less than or equal to 80 years old
2. Pathological diagnosis of rectal adenocarcinoma by colonoscopy biopsy
3. The distance between the tumor and the anal margin diagnosed by colonoscopy and pelvic MRI before operation is less than or equal to 15cm
4. No distant metastasis (including pelvic cavity, peritoneum, liver, lung, brain, bone, distant lymph node metastasis, etc.) is judged by ultrasound, CT, PET-CT, etc
5. No local complications before operation (no obstruction, incomplete obstruction, no massive active bleeding, no perforation, abscess formation, no local invasion)
6. Robot surgery
7. Voluntary participation and signing of informed consent

Exclusion Criteria:

1. Previous history of malignant colorectal tumors
2. Simultaneous diagnosis of multiple primary colorectal tumors
3. Those who have performed abdominal and pelvic surgery for many times or have extensive abdominal adhesions
4. Patients with familial adenomatous polyposis, Lynch syndrome associated rectal cancer, and inflammatory bowel disease at active stage
5. Diagnosis of other malignant tumors in recent 5 years
6. ASA grade ≥ IV and/or ECOG physical status score ≥ 2
7. Patients with severe liver and kidney function, heart and lung function, blood coagulation dysfunction or combined with severe basic diseases can not tolerate surgery
8. Preventive ileostomy
9. Patients undergoing combined abdominal and perineal resection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Incidence of anastomotic complications | 1 month after surgery
  Anastomotic leakage and anastomotic bleeding

SECONDARY OUTCOMES:
The number of stapler cartridges required for rectal transection | 1 month after surgery
  number per each surgery
operative time | 1 month after surgery
  minute
operative blood loss | 1 month after surgery
  milliliter
Time to first flatus | 1 month after surgery
  days
Postoperative length of stay | 1 month after surgery
  days
Distal resection margin | 1 month after surgery
  centimeter
proximal resection margin | 1 month after surgery
  centimeter

CONTACTS AND LOCATIONS:
Overall Officials: li taiyuan, doctor, Study Chair — The First Affiliated Hospital of Nanchang University
Locations (1):
- Taiyuan li, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No